CLINICAL TRIAL: NCT00000928
Title: Phase I Trial of an Intervention to Increase Condom Use by HIV-Discordant Couples
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HIVNET 013
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Sexual Partners; Condoms; Counseling
MeSH Terms: conditions — HIV Infections

ARMS (1):
- A (Experimental): All study participants
  Interventions: Behavioral: Group counseling intervention

INTERVENTIONS:
Behavioral: Group counseling intervention — Participants will engage in a multi-session group-based condom promotion program for approximately 12 months

SUMMARY:
To assess the acceptability of and participation in a group counseling intervention, including an assessment of willingness to disclose serostatus to a regular sexual partner and the willingness of that partner to participate. To evaluate the profile of adverse experiences (social, psychological, and physical harms) of individuals resulting from participation in counseling and testing and attempts to initiate condom use within a stable HIV serodiscordant partnership. To assess the potential for the intervention to result in increased condom use among stable sexual partners.

There is a significant risk of HIV transmission to HIV-uninfected partners in HIV-discordant couples. While condom use has been a major component of most AIDS prevention programs since the mid-1980s, there has been little emphasis on promoting condom use within stable partnerships. The most effective way to promote condom use among discordant couples remains largely unknown.

DETAILED DESCRIPTION:
There is a significant risk of HIV transmission to HIV-uninfected partners in HIV-discordant couples. While condom use has been a major component of most AIDS prevention programs since the mid-1980s, there has been little emphasis on promoting condom use within stable partnerships. The most effective way to promote condom use among discordant couples remains largely unknown.

A pilot study to assess the acceptability of intervention precedes the main study. The Phase I study recruits 15 HIV-infected men and 15 HIV-infected women and their partners at each of three sites (India, Thailand, and Uganda). Volunteers participate in a multi-session group-based condom promotion program for approximately 12 months. Couples are organized into small groups consisting of 4 to 6 couples per group. Each group meets for a total of 4 sessions within a 2- to 4-week period. Follow-up interviews are conducted at Months 1 and 3 following completion of the intervention.

ELIGIBILITY:
Inclusion Criteria

Volunteers must be:

* HIV-positive through HIVNET testing or HIV-seronegative by EIA.
* Presently in a sexual relationship of at least 6 months duration with the intention to remain with this partner for the duration of the study.
* Willing to identify and recruit this sexual partner to which he/she has disclosed or will disclose HIV serostatus.
* Willing to receive counseling and HIV testing (HIV-seronegative partners only).
* Willing to agree to be interviewed with their partner and individually.
* Willing to continue engaging in sex with their partner.
* Willing to participate in a couples-based condom promotion intervention.
* Willing and able to attend each scheduled intervention/follow-up study visit.

Exclusion Criteria

Volunteers with the following are excluded:

* History of domestic violence.
* Current consistent condom use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Primary Completion 1999-07 (Actual); Study Completion 1999-07 (Actual)

PRIMARY OUTCOMES:
Assess acceptability and participation | Throughout study
Assess the potential for the intervention to result in increased condom use among stable sexual partners | Throughout study

SECONDARY OUTCOMES:
Assessment of willingness to disclose serostatus to a regular sexual partner and the willingness of that partner to participate | Throughout study
Evaluation of adverse experiences (social, psychological, and physical harms) of individuals resulting from participation in counseling and testing | Throughout study
Evaluation of attempts to initiate condom use within a stable HIV serodiscordant partnership | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: David D. Celentano, Study Chair; Janet McGrath, Study Chair